CLINICAL TRIAL: NCT03265561
Title: Spinal Infection Management With Structural Allograft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Carlos A Acosta-Olivo, Prinicipal Investigator, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OR15-005
Record Dates: First submitted 2017-08-24; First posted 2017-08-29 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Bone Diseases, Infectious; Disease of Bone; Syndrome; Spine Infection; Allografts; Bone Graft; Complications, Fracture
MeSH Terms: conditions — Bone Diseases, Infectious; Bone Diseases; Syndrome; Fractures, Bone

STUDY DESIGN:
Intervention Model Description: Bone allograft group will receive bone structural allograft; Auto and allograft group will receive bone structural allograft plus spongy autograft.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone allograft group (Experimental): This participants will receive bone structural allograft management for vertebral reconstruction. All patients undergo surgical procedure to realize debridement of the lesion, and the application of allograft without autograft.
  Interventions: Device: Bone allograft
- Bone auto and allograft group (Active Comparator): This participants will receive bone structural allograft plus spongy autograft management for vertebral reconstruction. All patients undergo surgical procedure.
  Interventions: Device: Bone auto and allograft group

INTERVENTIONS:
Device: Bone allograft — All patients will undergo the same surgical procedure consisting of open surgery, more debridement of infected and devitalized tissue, as well as corresponding bone resection. For the identification of the microorganism, biopsies will be performed by puncture guided by CAT and / or fluoroscopy, and culture and antibiogram will be performed in case of not obtaining enough material for this, at the time of the surgery samples will be sent to perform the same procedure. We will use the appropriate antibiotics, according to infecting microorganism and result of antibiogram. We will include patients with infections with gram positive and negative microorganisms only. This patients will go stabilized with bone allograft only.
  Arms: Bone allograft group
Device: Bone auto and allograft group — All patients will undergo the same surgical procedure consisting of open surgery, more debridement of infected and devitalized tissue, as well as corresponding bone resection. For the identification of the microorganism, biopsies will be performed by puncture guided by CAT and / or fluoroscopy, and culture and antibiogram will be performed in case of not obtaining enough material for this, at the time of the surgery samples will be sent to perform the same procedure. We will use the appropriate antibiotics, according to infecting microorganism and result of antibiogram. We will include patients with infections with gram positive and negative microorganisms only. This patients will go stabilized with bone autograft plus bone allograft
  Arms: Bone auto and allograft group

SUMMARY:
Background. Bone infections can involve the vertebral column, intervertebral disc space, spinal canal and soft tissues, can generate neurological deficit in addition to the destruction of the bone that causes functional disability. Vertebral osteomyelitis is the most frequent, affecting 2 to 7 patients per 100,000 habitants. Management is bone debridement and bone reconstruction.

Objective. Demonstrate that the use of bone allograft is a functional method to stabilize the spine after a bone spinal infection Material and methods. Patients with vertebral bone destruction are included in two groups. Bone allograft group will receive bone structural allograft; Auto and allograft group will receive bone structural allograft plus autograft. The bone reconstruction will be performed in a one-time surgical procedure. Bone consolidation, pain, functionality, and spine deformity will be evaluated.

DETAILED DESCRIPTION:
Spinal bone infections can involve the bone vertebra, intervertebral disc space, spinal canal and soft tissues. It generate neurological deficit in addition to the destruction of the bone that causes functional disability and significant pain (Colmenero 1997). Spinal infections include discitis, osteomyelitis, epidural abscesses, meningitis, subdural empyema, and abscesses of the spinal cord (An, 2006). Only discitis and osteomyelitis can occur together (Skaf, 2010). Vertebral osteomyelitis is the most frequent, affecting 2 to 7 patients per 100,000 habitants (Bhavan, 2010; Grammatico 2003).

Pathogenic organisms reach the column by hematogenous pathway, arterial pathways (Batson's plexus) or by direct inoculation, due to a diagnostic or therapeutic intervention (Skaf, 2010). The natural history of pyogenic vertebral infections involves an infectious source or an incident followed by a period of intense pain, with or without generalized significant sepsis. Neurological deficit is caused by: [1] direct extension of the infection in the form of an abscess or bacterial communication with the spinal canal to the neural elements or [2] secondary compression of a pathological fracture as a result of bone softening. (Campbell´s, 2013).

Early diagnosis and treatment are essential for optimal outcomes (Weisz, 2000). The treatment goals may include eradicating the infection, relieving pain, preserving or restoring neurologic function, improving nutrition, and maintaining spinal stability (Tay, 2002). The aim of this study is to demonstrate that the use of bone allograft is a functional method to stabilize the spine after a bone spinal infection.

METHODS This study was approved by our Institutional Ethics and Research Committee. Patients with vertebral bone destruction are randomized included in two groups. Inclusion criteria: patients older than 18 years, any gender, pyogenic spinal infection with bone destruction and kyphotic deformity, without previous treatment of any kind, and Informed Consent signature. Exclusion criteria: patients with immunodeficiency, psychiatric disorders, patients with severe malnutrition, morbid obesity. Elimination criteria: failure to comply with follow-up time, patient's express request to leave the study. The bone reconstruction will be performed in a one-step surgical procedure. All participants will undergo the same surgical procedure consisting of open surgery, more debridement of infected and devitalized tissue, as well as corresponding bone resection. For the identification of the microorganism, biopsies will be performed guided by computed tomography (CT scan) and/or by fluoroscopy. A culture and antibiogram will be performed in case of not obtaining enough material for this, at the time of the surgery samples will be sent to perform the same procedure. The investigators will use the appropriate antibiotics, according to infecting microorganism and result of antibiogram, and patients with infections with gram positive and negative microorganisms only will be included. Bone consolidation, pain, functionality, and spinal deformity will be evaluated.

The investigators will perform evaluations at 8, 12, 16, 20 and 24 weeks, and a CT scan will be realized, to evaluated the bone consolidation, defined as the presence of continuous trabeculae between the bone graft and the vertebra, according to the next classification system. Type 1 definitive fusion; Type 2 uncertain fusion; Type 3 definitive pseudoarthrosis.

Statistical analysis. The results will be reported in contingency tables, frequencies, percentages, measures of central tendency and dispersion. Qualitative variables will be analyzed with the chi-square statistic and quantitative variables with t-test for independent samples with a significance level of 95% with their respective confidence intervals, or with non-parametric statistics if necessary. Using a formula for hypothesis testing and difference of two proportions or with the proportion of a reference value, with a value zα of 1.94 with a level of significance of 95% for a queue, and a value zβ of 1.20 with a power of 80 %, With a proportion for group 1 of 0.38 and for group 2 of 0.83 (Zdeblick, Ducker) a sample of 19 participants was obtained per group. Statistical analysis will be performed with IBM SPSS version 20 (SPSS, Inc., Armon, NY).

ELIGIBILITY:
Inclusion Criteria:

* pyogenic spinal infection with bone destruction and spinal deformity, without previous treatment of any kind and Informed Consent signature

Exclusion Criteria:

* immunodeficiency, psychiatric disorders, patients with severe malnutrition, morbid obesity

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Bone consolidation | Twelve months
  Radiography or CT scan will demonstrate bone graft consolidation

SECONDARY OUTCOMES:
Pain scale | Three months
  Visual Analogue Scale minimum 0 value = no pain; maximum 10 value= unsupportable pain
Oswestry Scale | Three months
  Oswestry Lumbar Pain Disability Scale
Degree of spinal deformity | Three months
  Radiographic measurement of Cobbs angle

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Acosta-Olivo, PhD, Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Universidad Autonoma de Nuevo Leon, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Colmenero JD, Jimenez-Mejias ME, Sanchez-Lora FJ, Reguera JM, Palomino-Nicas J, Martos F, Garcia de las Heras J, Pachon J. Pyogenic, tuberculous, and brucellar vertebral osteomyelitis: a descriptive and comparative study of 219 cases. Ann Rheum Dis. 1997 Dec;56(12):709-15. doi: 10.1136/ard.56.12.709. PMID 9496149
- [Background] An HS, Seldomridge JA. Spinal infections: diagnostic tests and imaging studies. Clin Orthop Relat Res. 2006 Mar;444:27-33. doi: 10.1097/01.blo.0000203452.36522.97. PMID 16523124
- [Background] Skaf GS, Domloj NT, Fehlings MG, Bouclaous CH, Sabbagh AS, Kanafani ZA, Kanj SS. Pyogenic spondylodiscitis: an overview. J Infect Public Health. 2010;3(1):5-16. doi: 10.1016/j.jiph.2010.01.001. Epub 2010 Feb 19. PMID 20701886
- [Background] Bhavan KP, Marschall J, Olsen MA, Fraser VJ, Wright NM, Warren DK. The epidemiology of hematogenous vertebral osteomyelitis: a cohort study in a tertiary care hospital. BMC Infect Dis. 2010 Jun 7;10:158. doi: 10.1186/1471-2334-10-158. PMID 20529294
- [Background] Grammatico L, Baron S, Rusch E, Lepage B, Surer N, Desenclos JC, Besnier JM. Epidemiology of vertebral osteomyelitis (VO) in France: analysis of hospital-discharge data 2002-2003. Epidemiol Infect. 2008 May;136(5):653-60. doi: 10.1017/S0950268807008850. Epub 2007 Jun 14. PMID 17568478
- [Background] Govender S. Spinal infections. J Bone Joint Surg Br. 2005 Nov;87(11):1454-8. doi: 10.1302/0301-620X.87B11.16294. No abstract available. PMID 16260656
- [Background] Reihsaus E, Waldbaur H, Seeling W. Spinal epidural abscess: a meta-analysis of 915 patients. Neurosurg Rev. 2000 Dec;23(4):175-204; discussion 205. doi: 10.1007/pl00011954. PMID 11153548
- [Background] Tay BK, Deckey J, Hu SS. Spinal infections. J Am Acad Orthop Surg. 2002 May-Jun;10(3):188-97. doi: 10.5435/00124635-200205000-00005. PMID 12041940
- [Background] Weisz RD, Errico TJ. Spinal infections. Diagnosis and treatment. Bull Hosp Jt Dis. 2000;59(1):40-6. PMID 10789037
- [Background] Mann S, Schutze M, Sola S, Piek J. Nonspecific pyogenic spondylodiscitis: clinical manifestations, surgical treatment, and outcome in 24 patients. Neurosurg Focus. 2004 Dec 15;17(6):E3. doi: 10.3171/foc.2004.17.6.3. PMID 15636573
- [Background] Sapico FL, Montgomerie JZ. Vertebral osteomyelitis. Infect Dis Clin North Am. 1990 Sep;4(3):539-50. PMID 2212605
- [Derived] Martinez-Gutierrez O, Pena-Martinez V, Camacho-Ortiz A, Vilchez-Cavazos F, Simental-Mendia M, Tamez-Mata Y, Acosta-Olivo C. Spondylodiscitis treated with freeze-dried bone allograft alone or combined with autograft: A randomized and blinded trial. J Orthop Surg (Hong Kong). 2021 May-Aug;29(2):23094990211019101. doi: 10.1177/23094990211019101. PMID 34041968